CLINICAL TRIAL: NCT01344148
Title: AIDS and Tuberculosis Co-infection Treatment Strategies Study of China.[ Eleven Fifth Key Research Grant From the Ministry of Science and Technology, the People's Republic of China]
Brief Title: Acquired Immunodeficiency Syndrome(AIDS) and Tuberculosis(Tb) Co-infection Treatment Strategies Study of China.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Lu Hongzhou, Shanghai Public Health Clinical Center Affiliated Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008ZX10001-008
Record Dates: First submitted 2010-09-14; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2008-08

CONDITIONS: AIDS
Keywords: Anti- TB; HAART; choice of the right moment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti- TB therapy HAART (Experimental)
  Interventions: Drug: INH RIF Rifb PZA EMB AZT 3TC D4T EFV

INTERVENTIONS:
Drug: INH RIF Rifb PZA EMB AZT 3TC D4T EFV — The first cohort study is the patients begin HAART after anti-TB therapy 2 weeks,and the second cohort is after 8 weeks begin HAART. Anti-TB therapy program is 2HREZ-4HRifb. And the first line of HAART plan is AZT+3TC+EFV and the second line plan is D4T+3TC+EFV.If begin with HAART and the RIF will change to Rifb.

SUMMARY:
To determine the best time to begin anti-HIV(Acquired Immunodeficiency Syndrome) treatment in individuals who co-infected with HIV and tuberculosis (Tb). This prospective, randomized study is being conducted on HIV/Tb co-infected patients in China to evaluate and compare the efficacy of antiretroviral therapy after 2 weeks TB treatment versus deferred ART initiated 8 weeks after initiation of TB treatment.

DETAILED DESCRIPTION:
Anti-Tb Therapy: 2HREZ-4HRifb(H:Isoniazid，R:Rifampicin，E:Ethambutol，Z：pyrazinamide，Rifb:Rifabutin) HAART: The first line was Zidovudine(AZT)+Lamivudine(3TC)+Efavirenz(EFV) and the second line is Stavudine(D4T)+3TC+EFV Study group one: after anti-TB therapy 2 weeks begin with High Active Antiretroviral Therapy(HAART); study group two: after anti-TB therapy 8 weeks begin with HAART. If begin with HAART and the H change with Rifb.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AIDS co-infected with TB CD4 T cell count lower than 350/ul Must be able to swallow tablets and finish the follow-up Sign the information consent form Chinese

Exclusion Criteria:

* Can not tolerance the therapy estimated by the doctor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 years
  In China TB is the main co-infected disease of AIDS patients. This study will give the evidence for make the HIV and TB Co-infected Patients therapy tactics of China. At first, the study will prove what is the best time for begin HAART after anti-TB therapy 2 weeks or 8 weeks. And anti-TB and HAART program will also be confirmed in this study. Overall this research will measure the HIV and TB co-infected patients clinical treatment safety and tolerability of China.

SECONDARY OUTCOMES:
Patients long-term survival. | 5 years
  The two groups will be follow up for more than five years and the long-term survival will be value.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hongzhou, MD. PhD, Study Chair — Shanghai Public Health Clinical Center Affliated to Fudan University China
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ji YJ, Liang PP, Shen JY, Sun JJ, Yang JY, Chen J, Qi TK, Wang ZY, Song W, Tang Y, Liu L, Zhang RF, Shen YZ, Lu HZ. Risk factors affecting the mortality of HIV-infected patients with pulmonary tuberculosis in the cART era: a retrospective cohort study in China. Infect Dis Poverty. 2018 Mar 24;7(1):25. doi: 10.1186/s40249-018-0405-8. PMID 29587840